CLINICAL TRIAL: NCT00685204
Title: A Phase II Study of Milataxel (TL139) Administered Orally in Patients With Malignant Mesothelioma
Brief Title: An Efficacy Study of Milataxel (TL139) Administered Orally for Malignant Mesothelioma
Acronym: TL139
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taxolog Inc. (Industry)
Responsible Party: Harvey Pass, M.D. Chief, Division of Thoracic Surgery and Thoracic Oncology, New York University Cancer Center
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: TL139204
Record Dates: First submitted 2008-05-21; First posted 2008-05-28 (Estimated); Last update posted 2008-05-28 (Estimated); Status verified 2008-05

CONDITIONS: Mesothelioma
MeSH Terms: conditions — Mesothelioma | interventions — MAC321

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): This is a non-random, multicenter, open label, single agent study. Patients with mailgnanat mesothelioma that has reccured or progressed following chemotherapy, and who qualify for this study, will receive oral milataxel.
  Interventions: Drug: Milataxel

INTERVENTIONS:
Drug: Milataxel — Milataxel is a liquid that is dosed orally at 60 mg/m2 on Day 1 of a 21 day cycle. If no toxicities of greater than Grade 1 severity occur, patients will receive 75 mg/m2 for the second and subsequent cycles.
  Other Names: TL139

SUMMARY:
Milataxel is a new taxane that may have several advantages over the currently available taxanes. The current study is designed to determine the response rate of oral Milataxel in patients with malignant Mesothelioma. The study specifically targets patients who have recurring or progressive disease following previous chemotherapy.

DETAILED DESCRIPTION:
This is a non-randomized, multicenter, open label, single agent phase II study. Patients with malignant mesothelioma that has recurred or progressed following chemotherapy, and who qualify for this study, will receive milataxel 60 mg/m2 orally on Day 1 of a 21 day cycle. If no toxicities of greater than Grade 1 severity occur, patients will receive 75 mg/m2 for the second and subsequent cycles. Patients will receive drug for a total of six cycles. Milataxel administration in excess of six cycles will be permitted at the discretion of the Investigator if patients have stable or responding disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed malignant mesothelioma for which they have received pemetrexed in combination with cisplatin as part of chemotherapeutic regimen.
* Prior cancer therapy with pemetrexed/cisplatin must have been completed at least 30 days prior to the first cycle of milataxel; prior radiotherapy (less than 25% of the bone marrow) must have been completed at least 30 days prior to study enrollment.
* Patients must have measurable disease by the Modified RECIST criteria
* Patients must have a life expectancy of at least 12 weeks and an ECOG performance status of 0, 1 or 2
* Patients must be 18 years of age.
* Patients must have adequate organ and system function.
* Patients must be able to comply with the protocol treatments and procedures.
* Patients with known brain metastases may be included in the study, providing they are clinically stable.
* Recovered from all acute toxicities caused by prior cancer therapies, except for alopecia.

Exclusion Criteria:

* Patients must not have received any other chemotherapeutic treatment for malignant mesothelioma other than pemetrexed and a platinum agent such as cisplatin.
* Patients with grade 2 or greater peripheral neuropathy.
* Prior cancer therapies not completed within 30 days prior to the first cycle of milataxel; radiotherapy completed less than 30 days prior to study enrollment; patients not recovered from radiation-related toxicities; patients receiving any concurrent anti-cancer therapy, including trastuzumab, bevacizumab or an investigational agent while on-study; patients with greater than 2 prior radiotherapy treatments.
* Patients with known sensitivity to alcohol.
* Patients with significant intercurrent illnesses.
* Patients with symptomatic CNS metastases.
* Patients who have had major surgery within the past 14 days.
* Patients who require or are likely to require any strong modifier of CYP450 activity to be taken prior to milataxel administration
* Patients who are receiving high dose steroids (more than a dexamethasone-equivalent dose of 4 mg per day).
* Patients with malabsorption syndrome, disease significantly affecting gastrointestinal function, or major resection of the stomach or small bowel that could affect absorption of the study drug.
* Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2008-03

PRIMARY OUTCOMES:
To determine the objective response rate of milataxel when given orally to previously treated patients with malignant mesothelioma.

SECONDARY OUTCOMES:
To evaluate time to progression, duration of tumor response and safety and tolerability of TL139 treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Harvey Pass, M.D., Principal Investigator — New York University Cancer Center
Locations (3):
- United States (3):
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - New York University Cancer Center, New York, New York